CLINICAL TRIAL: NCT02165553
Title: Acute Impact of Hibiscus Sabdariffa Calyces (HSC) Extract Consumption on Blood Pressure, Vascular Function and Other Cardiovascular Risk Factors
Brief Title: Impact of Hibiscus on Cardiovascular Disease Risk
Acronym: PHYTOVAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 13/40
Record Dates: First submitted 2014-06-01; First posted 2014-06-17 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Cardiovascular Diseases
Keywords: Hibiscus sabdariffa calyces; Blood Pressure; Vascular Function; Inflammation; Cardiometabolic risk markers; Systemic antioxidant capacity
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hibiscus sabdariffa calyces extract as a cold drink (Experimental): Subjects are asked to consume 250 ml of Hibiscus calyces drink after a high fat breakfast
  Interventions: Dietary Supplement: Hibiscus sabdariffa calyces extract as a cold drink
- Water (Placebo Comparator): Subjects are asked to consume 250 ml of water after a high fat breakfast
  Interventions: Dietary Supplement: Hibiscus sabdariffa calyces extract as a cold drink

INTERVENTIONS:
Dietary Supplement: Hibiscus sabdariffa calyces extract as a cold drink
  Other Names: Hibiscus flower tea; Hibiscus tea; Roselle

SUMMARY:
Hibiscus sabdariffa calyces (HSC) extract is consumed in different parts of the world as a cold or hot drink and is available in the United Kingdom (UK) markets in different forms including tea bags. There is preliminary data that support the hypothesis that HSC extract consumption has beneficial effect on blood vessel health and blood pressure reduction. Hypertension, vascular dysfunction, inflammation and lipid abnormalities are all key modifiable risk factors of cardiovascular diseases (CVD), the leading causes of death throughout the world. In the PHYTOVAS (PHYTOchemicals and VAScular Function) study the effect of the acute consumption a potentially bioactive food extracts: Hibiscus sabdariffa calyces (HSC) compared with a matched control (water) on blood pressure and blood vessels function will be investigated after a high - fat mixed meal. This is with a view to determining the impacts of the extract on postprandial (after meal) blood pressure and other CVD risk factors. Results from the PHYTOVAS study could lead to identification of more dietary approaches that will contribute to CVD risk prevention and management.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 30 - 65 years
* 1 to 10 % Cardiovascular disease risk in 10 years
* Not taking blood pressure medication
* Not having liver or kidney disease
* Not anaemic
* A signed consent form

Exclusion Criteria:

* Female
* <30 or > 65 years
* <1 or >10 % Cardiovascular disease risk in 10 years
* Taking blood pressure medication
* Having liver or kidney disease
* Anaemic
* Lack of signing consent form
* Vegan
* Individual with food allergy
* Sufferers of chronic illness

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in baseline and hourly blood pressure | Baseline, hourly 4 times post baseline and then hourly for twelve hours at night

SECONDARY OUTCOMES:
Change in Flow Mediated Vasodilation | Baseline, 2 and 4 hours post treatment
Change in blood lipids profile | Baseline and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4 hours post treatment
Change in Inflammatory marker: C - reactive protein (CRP) | Baseline and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4 hours post treatment
Change in plasma nitric oxide level | Baseline and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4 hours post treatment
Change in serum total antioxidant capacity | Baseline and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4 hours post treatment
Changes in serum or plasma glucose and insulin levels | Baseline and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4 hours post treatment

OTHER OUTCOMES:
Change in arterial stiffness measured by Pulse Wave Analysis (PWA) | Baseline, 2 and 4 hours post treatment
Pharmacokinetics of plasma anthocyanins and phenolic acids measured as Area Under the Concentration - Time Curve (AUC 0 - 4 hours for plasma) | Baseline and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4 hours post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Julie A. Lovegrove, BSc, PhD, RNutr, Principal Investigator — University of Reading; Jeremy P.E. Spencer, B.Sc, PhD, Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, University of Reading,, Reading, Berkshire, United Kingdom